CLINICAL TRIAL: NCT01818141
Title: An Open-label, Randomized Study to Assess Inhibition of Spore Production in Patients With Clostridium Difficile Infections: Fidaxomicin Versus Vancomycin
Brief Title: Study to Assess Inhibition of Spore Production in Patients With C. Difficile Infections: Fidaxomicin Versus Vancomycin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: Optimer Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NICO003785HE
Record Dates: First submitted 2013-03-19; First posted 2013-03-26 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-05

CONDITIONS: Clostridium Difficile Infection
MeSH Terms: conditions — Clostridium Infections | interventions — Vancomycin; Fidaxomicin

STUDY DESIGN:
Masking Description: Open-label
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fidaxomicin (Active Comparator): Fidaxomicin 200mg by mouth every 12 hours for 10 days
  Interventions: Drug: Fidaxomicin
- Vancomycin (Active Comparator): Vancomycin 125mg by mouth every 6 hours for 10 days
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Vancomycin — Vancomycin 125mg by mouth every 6 hours for 10 days
  Other Names: Vancomycin 125mg by mouth every 6 hours for 10 days
  Arms: Vancomycin
Drug: Fidaxomicin — Fidaxomicin 200mg by mouth every 12 hours for 10 days
  Other Names: Fidaxomicin 200mg by mouth every 12 hours for 10 days
  Arms: Fidaxomicin

SUMMARY:
The purpose of this study is to compare number of vegetative cells and spores in stool over time for fidaxomicin or vancomycin in patients diagnosed with their first episode of C. difficile infection.

DETAILED DESCRIPTION:
The purpose of this study is to:

* Compare quantitatively the number of vegetative cells in stool over time for fidaxomicin or vancomycin in patients diagnosed with their first episode of C. difficile infection
* Compare quantitatively the number of spores in the stool over time for patients presenting with their first episode of C. difficile infection having been treated with either fidaxomicin or vancomycin.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and above
* First diagnosis of C. difficile infection
* Treatment for C. difficile infection less than 24 hours
* Female subjects must be nonpregnant, nonlactating, and either postmenopausal for at least 1 year, surgically sterile (i.e., documented tubal ligation or hysterectomy) for at least 90 days, abstinent, or agree to use 1 of the following forms of contraception from the time of signing the Informed Consent form (ICF) until 30 days after leaving the study site: a nonhormonal intrauterine device (IUD) with spermicide, female condom with spermicide, contraceptive sponge with spermicide, diaphragm with spermicide, cervical cap with spermicide, a male sexual partner who agrees to use a male condom with spermicide, or a sterile sexual partner.

Exclusion Criteria:

* History of hypersensitivity to fidaxomicin or vancomycin
* Pregnant or breast-feeding
* Active treatment with other therapies with activity against C. difficile
* Receiving any peristaltic agents
* Medical history including ulcerative colitis or Chron's disease
* Ordered to be nothing by mouth or cannot swallow the study medication
* Participation in another clinical research study utilizing pharmacological treatment within 1 month or five half-lives of the medication whichever is longer
* Any other reason felt by the investigator to potentially affect the outcomes of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-10-17 (Actual); Primary Completion 2014-12-15 (Actual); Study Completion 2014-12-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

REFERENCES:
- [Result] Housman ST, Thabit AK, Kuti JL, Quintiliani R, Nicolau DP. Assessment of Clostridium difficile Burden in Patients Over Time With First Episode Infection Following Fidaxomicin or Vancomycin. Infect Control Hosp Epidemiol. 2016 Feb;37(2):215-8. doi: 10.1017/ice.2015.270. Epub 2015 Nov 23. PMID 26592763

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fidaxomicin | Vancomycin
Started | 18 | 16
Completed | 15 | 13
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 2 | 0
Not completed — No baseline C.diff colonies | 1 | 1
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fidaxomicin | Vancomycin | Total
Number analyzed (Participants) | 18 | 16 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (15) | 66 (15) | 67 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 7 | 7 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 16 | 15 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 18 | 16 | 34
Baseline total colony forming units (CFU) [Mean (Standard Deviation); unit: log10 CFU/g stool] — Total colony forming units (CFU) of Clostridium difficile per patient at baseline. This is the addition of vegetative cell counts and spore cell counts.
  log10 CFU/g stool | 5.41 (1.72) | 4.96 (1.81) | 5.19 (1.80)
Baseline spores CFU [Mean (Standard Deviation); unit: log10 CFU/g stool] — The count (colony forming units, CFU) of Clostridium difficile spores at baseline stool.
  log10 CFU/g stool | 5.00 (1.44) | 4.87 (1.43) | 4.94 (1.47)
Baseline vegetative cells CFU [Mean (Standard Deviation); unit: log10 CFU/g stool] — Count (colony forming units, CFU) of vegetative Clostridium difficile in baseline stool.
  log10 CFU/g stool | 4.23 (2.39) | 4.22 (2.1) | 4.23 (2.30)

OUTCOME MEASURES:

1. Primary Outcome: C. Difficile Spore Reduction of at Least 2 Log 10 Colony Forming Units (CFU)/g of Stool
Description: The number and percentage of patients who achieved at least 2 log10 colony forming units (CFU)/g of stool reductions of Clostridium difficile spores from baseline by the end of therapy (days 10-13).
Time Frame: day 10-13
Measure: Count of Participants; unit: Participants
Arm/Group | Fidaxomicin | Vancomycin
Number analyzed (Participants) | 12 | 9
Participants | 11 | 6

2. Primary Outcome: C. Difficile Vegetative Cell Reduction of at Least 2 Log 10 Colony Forming Units (CFU)/g of Stool
Description: The number and percentage of patients who achieved at least 2 log10 CFU/g of stool reductions of Clostridium difficile vegetative cells from baseline by the end of therapy (days 10-13)
Time Frame: day 10-13
Measure: Count of Participants; unit: Participants
Arm/Group | Fidaxomicin | Vancomycin
Number analyzed (Participants) | 7 | 5
Participants | 4 | 5

ADVERSE EVENTS:
Arm/Group | Fidaxomicin | Vancomycin
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/16
Other Adverse Events (participants affected / at risk) | 0/18 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No